CLINICAL TRIAL: NCT05532761
Title: Multidimensional Assessment of Quality of Life, Social and Professional Life and Care Utilization in Patients With Diffuse Large Cell B-cell Lymphoma Treated With CAR-T Cells
Acronym: QUALITOP CAR-T
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0430
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL); CAR-T Cells Treatment
Keywords: Diffuse large B-cell lymphoma (DLBCL); CAR-T cells; Quality of life; Real-life
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diffuse lare B cells lymphoma: Diffuse large B cells lymphoma patients eligibles for CAR-T cells therapy
  Interventions: Other: self-administered questionnaires

INTERVENTIONS:
Other: self-administered questionnaires — In order to describe the experience of CAR-T cell therapy of DLBCL patients, a pharmaceutical follow-up is carried out the day before the injection (baseline) and at 1, 3, 6, 9, 12 and 18 months. These follow-ups consist of interviews with the patient and the delivery of self-administered questionnaires. The interviews will investigate drug consumption, the use of self-medication and complementary alternative therapies and the adverse effects of interest. The self-questionnaires will focus on exploring multidimensional quality of life, social and professional life, anxiety-depression or uncertainty tolerance through internationally validated questionnaires.
  No supplementary visits will be needed : interviews with the research team will occur at the end of hematologic consultations.

SUMMARY:
Immunotherapy became in recent years a major innovation in the care of cancer patients, with unprecedented improvement in complete response and survival, particularly in hematological cancers. Since 2018, patients with relapsed or refractory lymphoma can benefit from immunotherapy based on CAR-T cells (Chimeric Antigenic Receptor - T cells), drugs derived from gene therapy and products from the patient's own T cells. The efficacy of these drugs, their development in more and more indications and in continuous earlier lines of treatment, their unprecedented adverse effects and their very high cost justify the search for predictive factors of efficacy and tolerance in order to optimize their use and benefit the greatest number of eligible patients. A better understanding of quality of life and its determinants in patients who received CAR-T cells could play a major role in predicting efficacy and tolerance. Quality of life data have indeed been deemed insufficient in phase 1-2 trials which have demonstrated the benefit of CAR-T cells in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) in 3rd line of treatment or more and led to obtaining their marketing authorization. It is therefore necessary to assess the quality of life of patients treated in routine care with CAR-T cells. The European Qualitop project aims, from self-questionnaires, to explore the quality of life during the 2 years following the initiation of immunotherapy with a multidimensional approach integrating genetic factors, lifestyle habits and psychosocial determinants of patients. In this context, the Qualitop CAR-T study is a prospective non-comparative real-life study aimed at describing the multidimensional quality of life, its psychosocial determinants and drug consumption in patients with relapsed or refractory DLBCL treated with CAR -T cells.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* eligible for treatment with CAR-Tcells (outside a clinical trial) in an indication of diffuse large B-cell lymphoma for which treatment with CAR-Tcells is scheduled
* follow-up in the Hematology department of the Hospices Civils de Lyon (Pr. Hervé Ghesquières)
* having given their non-objection to participate in the study.

Exclusion Criteria:

* Adults subject to a measure of legal protection (curatorship, guardianship)
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care and persons admitted to a health or social establishment
* People with a major psychiatric disorder likely to hinder the conduct of the study, in the opinion of the investigator
* Not fluent in French-
* simultaneous participation in another research involving the human person, except if it is a study falling within category 3 of the Jardé Law which does not call into question the follow-up of patients in the present study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse large cell B-cell lymphoma followed in the hematology department of Pr GUESQUIERES (Pierre-Bénite, France) whose treatment with CAR-T cells is planned will be offered participation in the QUALITOP CAR-T study.
  The number of patients with DLBCL benefiting annually from treatment with CAR-T cells in hematologic department is around 55.
  The number of subjects to be included, estimated at 30 patients over one year, is therefore compatible with the recruitment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change of mean score of FACT-Lym (Functional Assessment of Cancer Therapy - Lymphoma) quality of life | Baseline (day before chemotherapy of lymphodepletion), Month1, 3, 6, 9, 12 and 18 after injection of CAR-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Service pharmaceutique, Hospices Civils de Lyon - Groupement Hospitalier Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No